CLINICAL TRIAL: NCT06024811
Title: Investigation of the Effect of Supporting Nursing Care Provided in Line With Evidence-Based Practices During Intrapartum Period
Brief Title: Investigation of the Effect of Supporting Nursing Care Provided in Line With During Intrapartum Period
Acronym: Support
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Esra Cevik, Assist Prof., Balikesir University
Other Study IDs: Balikesir
Record Dates: First submitted 2023-07-25; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Delivery;Breech;Stillbirth
Keywords: supportive nursing care; state anxiety.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intervention: Pregnant women over 18 years of age, with cervical dilatation 3 cm or more, planned for spontaneous vaginal delivery, term and singleton pregnancy, who speak Turkish, who did not have language communication problems, and who voluntarily agreed to participate in the study were included.
  Pregnant women in the intervention and control groups were randomized using the "www.random.org website" on the computer (intervention=56 control= 56).Intervention and control groups were randomized according to some basic variables (age group, education level, body mass index, number of births and pregnancies, participation in prenatal preparation classes) considering the literature .
  Interventions: Behavioral: supporting nursing care
- control: Pregnant women over 18 years of age, with cervical dilatation 3 cm or more, planned for spontaneous vaginal delivery, term and singleton pregnancy, who speak Turkish, who did not have language communication problems, and who voluntarily agreed to participate in the study were included.
  During the data collection period of the study, 313 women were evaluated according to the inclusion and exclusion criteria. Women who did not meet the inclusion criteria (n=198) and refused to participate in the study (n=3) were not included in the study sample. Pregnant women in the intervention and control groups were randomized using the "www.random.org website" on the computer (intervention=56 control= 56).Intervention and control groups were randomized according to some basic variables (age group, education level, body mass index, number of births and pregnancies, participation in prenatal preparation classes) considering the literature (Taghenijad et al. 2010; Erdogan et al. 2017).

INTERVENTIONS:
Behavioral: supporting nursing care — Supportive nursing care was applied during the intrapartum period. Latent Active Transition phase,birt, postpartum period
  Other Names: Supportive nursing care practices in the latent phase Types of supportive care Physical Emotional Informational Advocacy Partner
  Groups: intervention

SUMMARY:
Aim: The aim of the research was to examine the effect of supportive nursing care provided in line with evidence-based practices during the intrapartum period.

DETAILED DESCRIPTION:
Methods Design and Settings This study with intervention-control group, randomized and intervention type was carried out in a hospital in Balikesir, located in the west of Turkiye.

Hypotheses Hypothesis 1: Supportive nursing care provided in line with evidence-based practices during the intrapartum period has an effect on the state anxiety level of women.

Hypothesis 2: Supportive nursing care provided in line with evidence-based practices during the intrapartum period has an effect on perceived labor pain.

Hypothesis 3: Supportive nursing care provided in the intrapartum period in line with evidence-based practices has an effect on the duration on birth.

Hypothesis 4: Supportive nursing care provided in line with evidence-based practices in the intrapartum period has an effect on maternal satisfaction.

Universe and sample of the research

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years of age,
* with cervical dilatation 3 cm or more,
* Planned for spontaneous vaginal delivery,
* Term and singleton pregnancy,
* Who speak Turkish, who did not have language communication problems,
* Who voluntarily agreed to participate in the study were included

Exclusion Criteria:

* Pregnant women with head-pelvis incompatibility
* Those who gave birth by cesarean section before
* Pregnant women planned for cesarean delivery
* Pregnant women with any systemic disease (Diabetes mellitus, hypertension, etc.)
* Pregnant women who develop fetal distress or hypoxia during labor)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women over 18 years of age.
Study Population: The universe of the research consisted of pregnant women who applied to the delivery unit of a hospital to give birth in Balıkesir, Turkiye. A total of 4634 deliveries took place in this hospital in 2019, of which 2315 were normal deliveries. (https://balikesirism.saglik.gov.tr/ accessed on 2021 Aug 18). The sample size in the study was calculated with the G*power 3.1.9.2 program. Since the scores will be compared in the two dependent groups before and after the intervention, the minimum sample size was calculated as 54, 27 people in each group, based on the two-way hypothesis, 5% type I error, 0.50 Cohen's effect size, and 95% power
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
positive birth | 2020-2021
  The positive birth highlights the importance of woman-centred care to optimize the experience of labour and childbirth for women and their babies through a holistic, human rights-based approach.

CONTACTS AND LOCATIONS:
Overall Officials: ESRA ÇEVİK, Principal Investigator — https://akademik.yok.gov.tr/AkademikArama/view/viewAuthor.jsp
Locations (1):
- Balıkesir University, Balıkesir, Altıeylül, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett SJ, Stark MA. Factors associated with labor support behaviors of nurses. J Perinat Educ. 2010 Winter;19(1):12-8. doi: 10.1624/105812410X481528. PMID 21197128
- [Background] Bohren MA, Hofmeyr GJ, Sakala C, Fukuzawa RK, Cuthbert A. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2017 Jul 6;7(7):CD003766. doi: 10.1002/14651858.CD003766.pub6. PMID 28681500
- [Background] Cicek S, Basar F. The effects of breathing techniques training on the duration of labor and anxiety levels of pregnant women. Complement Ther Clin Pract. 2017 Nov;29:213-219. doi: 10.1016/j.ctcp.2017.10.006. Epub 2017 Oct 18. PMID 29122264
- [Background] Debeb Sendekie A, Belay MA, Ayalew Yimer S, Degu Ayele A. Evidence-Based Intrapartum Practice and Associated Factors Among Obstetric Care Providers Working in Public Hospitals of South Wollo Zone North-Central Ethiopia: An Institutional-Based Cross-Sectional Study. Int J Womens Health. 2022 May 19;14:719-730. doi: 10.2147/IJWH.S351795. eCollection 2022. PMID 35615384
- [Background] Gams B, Neerland C, Kennedy S. Reducing Primary Cesareans: An Innovative Multipronged Approach to Supporting Physiologic Labor and Vaginal Birth. J Perinat Neonatal Nurs. 2019 Jan/Mar;33(1):52-60. doi: 10.1097/JPN.0000000000000378. PMID 30676462
- [Background] Silva Gallo RB, Santana LS, Jorge Ferreira CH, Marcolin AC, Polineto OB, Duarte G, Quintana SM. Massage reduced severity of pain during labour: a randomised trial. J Physiother. 2013 Jun;59(2):109-16. doi: 10.1016/S1836-9553(13)70163-2. PMID 23663796
- [Background] Hodnett ED, Gates S, Hofmeyr GJ, Sakala C. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003766. doi: 10.1002/14651858.CD003766.pub2. PMID 17636733
- [Background] Hodnett ED, Gates S, Hofmeyr GJ, Sakala C. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2012 Oct 17;10:CD003766. doi: 10.1002/14651858.CD003766.pub4. PMID 23076901
- [Background] Kobayashi S, Hanada N, Matsuzaki M, Takehara K, Ota E, Sasaki H, Nagata C, Mori R. Assessment and support during early labour for improving birth outcomes. Cochrane Database Syst Rev. 2017 Apr 20;4(4):CD011516. doi: 10.1002/14651858.CD011516.pub2. PMID 28426160
- [Background] Nikula P, Laukkala H, Polkki T. Mothers' Perceptions of Labor Support. MCN Am J Matern Child Nurs. 2015 Nov-Dec;40(6):373-80. doi: 10.1097/NMC.0000000000000190. PMID 26275315
- [Background] Mortazavi SH, Khaki S, Moradi R, Heidari K, Vasegh Rahimparvar SF. Effects of massage therapy and presence of attendant on pain, anxiety and satisfaction during labor. Arch Gynecol Obstet. 2012 Jul;286(1):19-23. doi: 10.1007/s00404-012-2227-4. Epub 2012 Jan 21. PMID 22271239
- [Background] Smith CA, Levett KM, Collins CT, Dahlen HG, Ee CC, Suganuma M. Massage, reflexology and other manual methods for pain management in labour. Cochrane Database Syst Rev. 2018 Mar 28;3(3):CD009290. doi: 10.1002/14651858.CD009290.pub3. PMID 29589380
- [Background] Weeks F, Pantoja L, Ortiz J, Foster J, Cavada G, Binfa L. Labor and Birth Care Satisfaction Associated With Medical Interventions and Accompaniment During Labor Among Chilean Women. J Midwifery Womens Health. 2017 Mar;62(2):196-203. doi: 10.1111/jmwh.12499. Epub 2016 Aug 20. PMID 27543442
- [Background] Wanyenze EW, Nalwadda GK, Byamugisha JK, Muwanguzi PA, Tumwesigye NM. Effect of Midwife-Provided Orientation of Birth Companions on Maternal Anxiety and Coping during Labor: A Stepped Wedge Cluster Randomized Control Trial in Eastern Uganda. Int J Environ Res Public Health. 2023 Jan 14;20(2):1549. doi: 10.3390/ijerph20021549. PMID 36674304
- [Result] Dai XW. [Scanning electron microscopy of gallstone matrix]. Zhonghua Wai Ke Za Zhi. 1983 Jun;21(6):326-7. No abstract available. Chinese. PMID 6641424